CLINICAL TRIAL: NCT04157608
Title: Evaluation of an Energy-Harvesting Mesofluidic Impulse Prosthesis (e-MIP) in Transtibial Prosthesis Users
Brief Title: Energy-Harvesting Mesofluidic Impulse Prosthesis: e-MIP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigational device under development
Sponsor: Orthocare Innovations, LLC (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 0309-02; 2R44HD080309 (NIH)
Record Dates: First submitted 2019-10-31; First posted 2019-11-08 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Transtibial Amputation; Artificial Limbs

STUDY DESIGN:
Intervention Model Description: Crossover clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Habitual Prosthesis (Active Comparator): Participant's existing baseline prescribed prosthesis
  Interventions: Device: Habitual Prosthesis
- e-MIP (Experimental): Experimental ankle-foot prosthesis
  Interventions: Device: Energy-Harvesting Mesofluidic Impulse Prosthesis

INTERVENTIONS:
Device: Habitual Prosthesis — Habitual baseline prosthesis prescribed by participant's clinician.
  Arms: Habitual Prosthesis
Device: Energy-Harvesting Mesofluidic Impulse Prosthesis — e-MIP is an experimental lower limb ankle-foot prosthesis.
  Arms: e-MIP

SUMMARY:
The purpose of this research is to validate the e-MIP design and function by testing the ability of e-MIP to harvest energy and return a sufficient amount of energy to assist the user during gait. The investigators will also evaluate whether prosthetic users are able to wear and use the e-MIP device long-term.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transtibial amputation
* At least twelve months post-amputation
* Currently walking on a prosthesis for at least one year
* Uses modular endoskeletal prosthetic components
* Has bilateral normal range of motion
* Ability to walk independently and for an extended length of time (walking ability of each individual will be assessed by the principal investigator or study prosthetist during the recruitment period)
* Ability to communicate individual perceptions
* Ability to provide informed consent

Exclusion Criteria:

* Confounding injury or musculoskeletal problem
* Pregnancy
* Lower limb peripheral neuropathy
* Symptomatic cardiovascular disease or chronic obstructive pulmonary disease
* Not able to read and understand English

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2022-07-10 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
Energy returned | After four weeks with Habitual Prosthesis
  The amount of energy returned at the ankle joint, calculated from ankle torque and angle sensors with respect to time.
Energy returned | After four weeks with e-MIP (system ON and system OFF)
  The amount of energy returned at the ankle joint, calculated from ankle torque and angle sensors with respect to time.

SECONDARY OUTCOMES:
Total Steps | After four weeks with Habitual Prosthesis
  The number of steps taken by the participant will be recorded over four weeks with a step activity monitor.
Total Steps | After four weeks with e-MIP (system ON and system OFF)
  The number of steps taken by the participant will be recorded over four weeks with a step activity monitor.
Step Rate | After four weeks with Habitual Prosthesis
  The speed of steps taken by the participant will be recorded over four weeks with a step activity monitor.
Step Rate | After four weeks with e-MIP (system ON and system OFF)
  The speed of steps taken by the participant will be recorded over four weeks with a step activity monitor.
Step Activity | After four weeks with Habitual Prosthesis
  The number of continuous steps taken by the participant will be recorded over four weeks with a step activity monitor.
Step Activity | After four weeks with e-MIP (system ON and system OFF)
  The number of continuous steps taken by the participant will be recorded over four weeks with a step activity monitor.
Prosthesis Evaluation Questionnaire | After four weeks with Habitual Prosthesis
  Responses to the psychometrically validated scales of the Prosthesis Evaluation Questionnaire for persons with limb loss, in order to understand the participant's perception of the prosthesis. Questionnaire scores range from 0 to 100. Higher scores indicate a better outcome.
Prosthesis Evaluation Questionnaire | After four weeks with e-MIP (system ON and system OFF)
  Responses to the psychometrically validated scales of the Prosthesis Evaluation Questionnaire for persons with limb loss, in order to understand the participant's perception of the prosthesis. Questionnaire scores range from 0 to 100. Higher scores indicate a better outcome.
Spatio-Temporal Gait Parameters | After four weeks with Habitual Prosthesis
  The spatio-temporal parameters of gait, such as walking speed, will be measured using motion analysis.
Spatio-Temporal Gait Parameters | After four weeks with e-MIP (system ON and system OFF)
  The spatio-temporal parameters of gait, such as walking speed, will be measured using motion analysis.
Kinematics during Gait | After four weeks with Habitual Prosthesis
  Kinematics such as hip, knee, and ankle joint angles will be measured using motion analysis.
Kinematics during Gait | After four weeks with e-MIP (system ON and system OFF)
  Kinematics such as hip, knee, and ankle joint angles will be measured using motion analysis.
Kinetics during Gait | After four weeks with Habitual Prosthesis
  Kinetics such as hip, knee, and ankle joint torques will be measured using motion analysis.
Kinetics during Gait | After four weeks with e-MIP (system ON and system OFF)
  Kinetics such as hip, knee, and ankle joint torques will be measured using motion analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Orthocare Innovations, LLC, Edmonds, Washington, United States

IPD SHARING:
Plan to Share IPD: No